CLINICAL TRIAL: NCT05949866
Title: Feasibility and Fidelity of a Gross Motor-based Physical Activity Intervention on Cognitive Variables in Preschool-age Children From Low Socioeconomic Backgrounds.
Brief Title: Feasibility and Fidelity of a Gross Motor-based Physical Activity Intervention on Cognition in Preschool-age Children
Acronym: P-MAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Sofiya Alhassan, Professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21HD108125-01A1 (NIH)
Record Dates: First submitted 2023-06-15; First posted 2023-07-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-03

CONDITIONS: Activity, Motor
Keywords: Physical activity; Gross motor skills; Train-the trainer model; Cognition
MeSH Terms: conditions — Motor Activity | interventions — Movement; Control Groups

STUDY DESIGN:
Intervention Model Description: Childcare centers will be randomized to either the treatment or the control intervention.
Who Masked: Outcomes Assessor
Masking Description: Data collectors (outcome assessors) collecting cognition outcome variables will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Movement and Cognition Intervention group (MAC) (Experimental): Movement and Cognition group is the behavioral treatment group.
  Interventions: Behavioral: Movement and Cognition Intervention Group
- Health Tracker group (Control) (Placebo Comparator): Health tracker group is the control group.
  Interventions: Behavioral: Health Tracker Group (Control Group)

INTERVENTIONS:
Behavioral: Movement and Cognition Intervention Group — Preschool centers assigned to the Movement and Cognition (MAC) group will receive the 6-month intervention, which will be implemented 4 days per week. To ensure consistency of intervention delivery, centers will be provided with the MAC modules on a bi-weekly basis. The MAC intervention will be implemented using a train-the-trainer (gradual release) model. This will be a gradual release model, in which interventionist will first serve as a co-provider and will eventually serve in a support role, as providers become primary implementers.
  The MAC intervention will consist of gross motor skill curriculum consists of 30 individual lesson plans. The number of days needed to instruct each lesson plan activities ranges between 3 to 5 days. In each lesson, specific instruction and activities are designed to teach fundamental movements (e.g., running, leaping, kicking, jumping, throwing, catching).
  Arms: Movement and Cognition Intervention group (MAC)
Behavioral: Health Tracker Group (Control Group) — Preschool centers assigned to the health tracker g group will be asked to maintain their usual daily schedule and to not participate in other physical activity programs during the 6-month intervention.
  Arms: Health Tracker group (Control)

SUMMARY:
The goal of this study will be to examine the implementation and preliminary efficacy of a teacher taught gross motor skill-based physical activity (PA) intervention on cognitive variables in low low socio-economic (SES) preschoolers. The movement and cognition intervention will be implemented for 4 days per week for 6 months. Primary outcome variables will be processed evaluation data. Secondary outcome variables will be changes in children's cognitive function (executive functions and memory), gross motor skills, and PA levels at baseline, 3- and 6-month.

DETAILED DESCRIPTION:
The goal of this study will be to examine the implementation and preliminary efficacy of a teacher taught gross motor skill-based physical activity (PA) intervention on cognition in low low socio-economic (SES) preschoolers. Low SES preschool centers (n=4) will be recruited and randomly assigned to either a Movement and Cognition (MAC) or a control group. From each preschool center, preschool-age children will be recruited to participate in their assigned center intervention. The MAC intervention will be implemented for 4 days per week for 6 months. The research team will train the preschool providers to implement the intervention. The control centers will be asked to maintain their usual preschool schedule. Primary outcome variables will be processed evaluation data [study fidelity (adherence, compliance, and integrity of study design), intervention dosage, acceptability, quality, adaptation], and will be assessed throughout the 6-month study. Secondary outcome variables will be changes in children's cognitive function (executive functions and memory), gross motor skills, and PA levels at baseline, 3- and 6-month. Aim 1 will examine the implementation of a 6-month teacher taught gross motor skill-based movement intervention in low SES preschoolers. Aim 2 will examine the preliminary efficacy of the MAC intervention on cognition, gross motor skills, and PA in preschoolers. For aim 2, the study will compare the outcome variables of interest between the MAC and the control group.

ELIGIBILITY:
All children within a childcare center will participate in center's assigned activities. However, children will be individually recruited to participate in the measurement portion of study.

Childcare center will be eligible for study if:

* They have at least 40 (preschool-age) children enrolled
* Have at least 2 full-day preschool classrooms
* Not concurrently participating in other physical activity or gross motor skills programs

Child will be eligible for measurement portion of the study and the parent component if she or he is

- 3 - 5 years old at baseline assessment

Children will be excluded from the measurement portion of the study if they:

* Have conditions limiting participation in gross motor skills or physical activity intervention or the assessment of physical activity
* Plan to move away from the Springfield, MA area within the next 6 months.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Implementation - Study fidelity | Through out the 6 months intervention
  Process evaluation data, specifically the study fidelity of the intervention, will be assessed.
  On 2 randomly selected days per week within the treatment preschool center classrooms, research staff members will directly observe the intervention and use a semi-structured questionnaire (created by research PI) to collect information on intervention study fidelity (are the intervention activities being implemented as designed). In addition, 1 day per week, research staff members will directly observe the control center and use a semi-structured questionnaire to assessment of control (CON) school activities.
Implementation - Quality | Through out the 6 months intervention
  This will be assessed how well intervention training was delivered to providers & research staff.
  On 2 randomly selected days per week within the treatment preschool center classrooms, research staff members will directly observe the intervention and use a semi-structured questionnaire (created by research PI) to collect information on intervention study fidelity (quality of the intervention implementation by classroom providers).
Implementation - Adaptation | Through out the 6 months intervention
  Weekly survey with researchers and providers during 6-month program at both Movement and Cognition (MAC) and control (CON) centers to determine if there was any modification to either the MAC or the CON program.
Implementation - Dose delivered | Through out the 6 months intervention
  Process evaluation data on how much of the intervention was delivered.
  This will be assessed using the weekly log of Movement and Cognition (MAC) implementation by research staff and childcare providers.
Implementation - Acceptability | Completion of 6 months intervention
  A semi-structured questionnaire with providers at the completion of 6-month intervention in the Movement and Cognition (MAC) group. This will address the acceptability and satisfaction of the overall program and the individual intervention components.
Implementation - Intervention intensity | Through out the 6 months intervention
  Process evaluation data on the intervention intensity.
  Children in both the Movement and Cognition (MAC) and control (CON) centers will be asked to wear the activity accelerometer on one random day per week to assess the intervention intensity.

SECONDARY OUTCOMES:
Change in preschoolers cognition | Baseline, 3-month and 6-month
  Preschoolers' cognition will be assessed using via the NIH Toolbox for Assessment of Neurological and Behavioral Function on an iPad.
Change in preschoolers' behavioral outcome | Baseline, 3-month and 6-month
  Preschoolers' behavioral outcome will be assessed with the Children's Behavior Questionnaire (Very Short Form).
Change in preschoolers' gross motor skills | Baseline, 3-month and 6-month
  Preschoolers' gross motor skills will be assessed with the Test of Gross Movement Development, 3rd edition (TGMD-3).
Change in preschoolers moderate-to-vigorous physical activity | Baseline, 3-month and 6-month
  Preschoolers physical activity will be assessed with accelerometers for 7 consecutive days at each time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Sofiya Alhassan, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States